CLINICAL TRIAL: NCT02856490
Title: A Pilot Study to Determine the Degree and Effectiveness of the Various Operating Modes of vSculpt on Enhancing Genital Blood Flow and Improving Quality of Life in Women Who Experience Sexual Dysfunction and Stress Incontinence
Brief Title: A Study to Measure the Degree and Effectiveness of the Various vSculpt Operating Modes
Status: Completed | Type: Interventional
Sponsor: Joylux, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JOY 1515-02
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2016-08

CONDITIONS: Sexual Dysfunction; Stress Incontinence
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (3):
- vSculpt with Vibration Only (Active Comparator): vSculpt genital device used in vibration mode only.
  Interventions: Device: vSculpt
- vSculpt with Vibration and Light (Active Comparator): vSculpt genital device used in vibration and light mode.
  Interventions: Device: vSculpt
- InTone Device (Active Comparator): InTone genital device using electric muscle stimulation only.
  Interventions: Device: InTone

INTERVENTIONS:
Device: vSculpt — A genital vibration device that operates in two modes, vibration only or vibration and light, to help tone and tighten pelvic floor muscles.
  Arms: vSculpt with Vibration Only; vSculpt with Vibration and Light
Device: InTone — A genital device using electric muscle stimulation to treat incontinence.
  Other Names: ApexM
  Arms: InTone Device

SUMMARY:
A pilot study to determine the degree and effectiveness of the various modes of vSculpt, an over-the-counter "OTC" medical device, on enhanced genital blood flow and improvement in quality of life in menopausal women who suffer sexual dysfunction and stress incontinence

DETAILED DESCRIPTION:
The primary aim of this study is to determine the degree and effectiveness of the various modes of vSculpt on enhanced genital blood flow with menopausal women who experience sexual dysfunction and stress incontinence as measured by temperature change in the genitalia immediately after initial and final treatment and an improvement in quality of life after using the vSculpt device over the course of four weeks. The secondary aim is to compare the differences in genital blood flow and improvement in quality of life of vSculpt's various modes against Intone, another over-the-counter "OTC" medical device that utilizes a different technology to treat stress incontinence and improve sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be female
* Female participants who are capable of giving informed consent
* Female participants who are menopausal who have not had a menses within one year, and are within the ages of 48 and 60
* Female participants who have had one or more vaginal births
* Female participants who are currently engaged in vaginal sexual intercourse with a partner
* Female participants who are presently experiencing bladder control issues either leakage, frequency or urgency
* Female participants who are presently experiencing pain during sexual intercourse

Exclusion Criteria:

* Female participants shall not have an active sexually transmitted disease and/or infection
* Female participants who are actively undergoing chemotherapy
* Female participants who are currently taking any cancer-related drugs
* Female participants who are breastfeeding or lactating
* Female participants who have a medical history of neurological disorders (e.g., multiple sclerosis, Parkinson's disease)
* Female participants with an active urinary tract infection (UTI)
* Female participants with active bladder stones
* Female participants with active bladder tumor(s)
* Females with prior laser or vaginal rejuvenation surgeries or treatments
* Females with a medical history of vaginal cancer or radiation or surgery with exception of related to childbirth
* Females with prior non-invasive treatments (estrogen cream) or pelvic floor physical therapy for the vaginal area/ pelvic floor in the past six month
* Females with a physical disability precluding her from holding a lithotomy for an hour
* Females who are homeless

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Flow as Measured by Temperature Change in the Genitalia Using Thermography Technology
Description: The primary outcomes assessed will be change in blood flow as measured by temperature change in Celsius in the genitalia using thermography technology.
Time Frame: Pre and post treatment at baseline and pre and post treatment at day 30
Measure: Mean (Standard Deviation); unit: Celsius degree
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Number analyzed (Participants) | 2 | 2 | 2
Celsius degree
  Baseline | -0.5 (0.7) | 1.8 (1.3) | -0.3 (0.7)
  30 Days Post Treatment | -0.2 (0.4) | 0 (2.0) | -0.8 (0.1)

2. Secondary Outcome: Patient Quality of Life as Measured by Female Sexual Function Index (FSFI) Scores at Baseline and 30 Days Post Treatment.
Description: Change in patient quality of life as measured by an improvement in Female Sexual Function Index (FSFI) scores at baseline and 30 days post treatment. The range being from 2 (minimum) to 36 (maximum), with maximum being better.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Number analyzed (Participants) | 2 | 2 | 2
units on a scale
  Baseline | 13.9 (1.1) | 21.6 (6.0) | 22.7 (8.3)
  30 Days Post | 19.0 (5.7) | 29.6 (2.3) | 22.3 (5.5)

3. Secondary Outcome: Patient Quality of Life as Measured by Female Sexual Distress Scores (FSDS) at Baseline and 30 Days Post Treatment.
Description: Change in patient quality of life as measured by an improvement in Female Sexual Distress Scores (FSDS) at baseline and 30 days post treatment. The range being from 0 (minimum) to 52 (maximum), with minimum being better.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Number analyzed (Participants) | 2 | 2 | 2
units on a scale
  Baseline | 25.5 (12.0) | 22.0 (5.7) | 11.0 (5.7)
  30 Days Post | 20.0 (5.7) | 19.5 (2.1) | 5.0 (2.8)

4. Secondary Outcome: Patient Quality of Life as Measured by the Urogenital Distress Inventory, Short Form (UDI-6)
Description: Change in patient quality of life as measured by an improvement in Urogenital Distress Inventory, Short Form (UDI-6) scores. The range being from 0 (minimum) to 100 (maximum), with minimum being better.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Number analyzed (Participants) | 2 | 2 | 2
units on a scale
  Baseline | 30.6 (3.9) | 72.2 (15.7) | 47.2 (27.5)
  30 Days Post | 33.3 (7.9) | 41.7 (19.6) | 36.1 (19.6)

5. Secondary Outcome: Patient Quality of Life as Measured by the Incontinence Impact Questionnaire, Short Form (IIQ-7)
Description: Change in patient quality of life as measured by an improvement in Incontinence Impact Questionnaire, Short Form (IIQ-7) scores. The range being from 0 (minimum) to 100 (maximum), with minimum being better.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
Number analyzed (Participants) | 2 | 2 | 2
units on a scale
  Baseline | 9.5 (13.5) | 47.6 (26.9) | 14.3 (20.2)
  30 Days Post | 9.5 (6.7) | 40.5 (43.8) | 2.4 (3.4)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | vSculpt With Vibration Only | vSculpt With Vibration and Light | InTone Device
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other